CLINICAL TRIAL: NCT06232993
Title: Comparative Evaluation of the Effects of Kinesio Tape and Occlusal Splint Use in the Management of Myofascial Pain in Children With Sleep Bruxism: A Randomized Controlled Trial
Brief Title: Management of Myofascial Pain in Children With Sleep Bruxism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University (Other)
Responsible Party: Principal Investigator, Kamile Nur Tozar, Dr, Adiyaman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Decision number:2022-4-2
Record Dates: First submitted 2023-10-13; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Bruxism
MeSH Terms: conditions — Bruxism | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- occlusal splint (Experimental): A 0.5 mm thick hard thermoplastic acrylic plate was adapted to the model in the laboratory and prepared to cover the occlusal, buccal, and lingual surfaces of the teeth
  Interventions: Other: Kinesio taping
- kinesio taping (Experimental): The tape was cut into 2 pieces of an 'I' shape, approximately 5 cm long and 2.5 cm wide, according to the instructions in the manual.
  Interventions: Other: Occlusal Splinting
- exercises (Experimental): Participants in the EG group performed the exercises twice a day, with 10 repetitions and 3 sets for 5 weeks.
  Interventions: Other: Exercises

INTERVENTIONS:
Other: Kinesio taping — Kinesio taping is a technique that involves the application of a special elastic tape to the skin to provide support to muscles and joints without restricting the body's range of motion. This method is designed to facilitate the body's natural healing process and improve muscle function while providing support and stability to muscles and joints. Kinesio tape is believed to help reduce pain, support muscles during movement, and aid in rehabilitation. It is commonly used in sports medicine and physical therapy to address a variety of musculoskeletal conditions and injuries.
  Arms: occlusal splint
Other: Occlusal Splinting — Occlusal splinting, also known as a bite guard or night guard, is a removable dental appliance typically made of plastic that is custom-fitted to a patient's upper or lower teeth. It is primarily used to address issues related to teeth grinding (bruxism) or temporomandibular joint (TMJ) disorders. The splint is designed to fit over the teeth, creating a barrier between the upper and lower teeth to prevent grinding and clenching during sleep. Occlusal splints aim to reduce the impact of bruxism on the teeth and jaw, alleviate associated pain, protect the teeth from wear, and promote relaxation of the jaw muscles.
  Arms: kinesio taping
Other: Exercises — For patients with bruxism, exercises can be beneficial in managing symptoms and promoting relaxation of the jaw muscles. These exercises aim to reduce the frequency and intensity of bruxism, alleviate associated pain, and improve overall jaw function and comfort. It's important for patients to consult with healthcare professionals to determine the most appropriate exercises for their individual needs.
  Arms: exercises

SUMMARY:
This study compared the effectiveness of Kinesio tape and occlusal splint application in improving sleep quality and reducing myofascial pain in children with sleep bruxism.

DETAILED DESCRIPTION:
Forty-seven pediatric patients with sleep bruxism symptoms were randomly assigned into 3 groups for treatment: Kinesio tape group (KT), Occlusal splint group (OS), and Exercise group (EG). The following assessments were made in all 3 groups, before the treatment and at the end of the 1st and 5th week: Wong-Baker Faces Pain Scale (WBFPS), measurement of maximum mouth opening, assessment of pressure pain threshold of the bilateral masseter and temporal muscles, and evaluation of temporal and masseter muscle thickness by ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-11 years [1] presented to the clinic and had at least one symptom of sleep bruxism,
* Children and parents who agreed to participate in the study,
* Children who have not been treated for sleep bruxism before,
* Children who can cooperate,
* Children without maxillofacial trauma.

Exclusion Criteria:

* • Children with psychiatric/neurological/systemic disorders,

  * Children with a history of allergies or asthma,
  * Children using orthodontic appliances,
  * Children taking any medication,
  * Children with dental abscess or fistula mouth,
  * Children using a fixed or removable placeholder appliance.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Wong-Baker Faces Pain Scale | Applied before, 1 week after, and 5 weeks after the treatment
  The Wong-Baker Faces Pain Scale is a pain assessment tool that uses a series of faces to help individuals, especially children, express the intensity of their pain. It consists of a line of faces ranging from a smiling face (indicating "no pain") to a face with a distressed expression (indicating "worst pain"). The person is asked to point to the face that best represents their level of pain, allowing healthcare providers to assess and understand the individual's pain experience, particularly in cases where verbal communication may be challenging.

CONTACTS AND LOCATIONS:
Overall Officials: Kamile N Tozar, Principal Investigator — Adıyaman U
Locations (1):
- Adiyaman Universty, Adıyaman, Turkey (Türkiye)